CLINICAL TRIAL: NCT06995118
Title: The Application of "HUAXI Hole 1" in Reverse-sequence Endoscopic Nipple-sparing Mastectomy With Direct-to-implant Breast Reconstruction: A National Multicenter, Open-Label, Randomized Controlled Trial (HUAXI-h-01)
Brief Title: The Application of "HUAXI Hole 1" in Reverse-sequence Endoscopic Nipple-sparing Mastectomy With Direct-to-implant Breast Reconstruction
Acronym: HUAXI-h-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Du Zhenggui (Other)
Collaborators: West China Tianfu Hospital, Sichuan University (Unknown); West China Fourth Hospital, Sichuan University (Unknown); The Fourth People's Hospital of Sichuan Province (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); The First Hospital of Jilin University (Other); Shanxi Bethune Hospital (Other); Chengdu Fifth People's Hospital (Other); Suzhou Municipal Hospital (Other); Taiyuan Central Hospital of Shanxi Medical University (Other); The People's Hospital of DAZU ，Chongqing (Unknown); Anyang City Tumor Hospital (Unknown); Mianyang Hospital of Traditional Chinese Medicine (Unknown); Sichuan Cancer Hospital and Research Institute (Other); Deyang People's Hospital (Other); Hunan University of Traditional Chinese Medicine (Other); The Affiliated Hospital of lnner Mongolia Medical University (Unknown); Guangzhou First People's Hospital (Other); Fujian Medical University Union Hospital (Other); Nanchang People's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Du Zhenggui, Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024(2591)
Record Dates: First submitted 2025-05-07; First posted 2025-05-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast Cancer; Endoscopic surgery; Nipple-sparing mastectomy; Minimal invasive surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HH-01 group (Experimental): Use 'HUAXI hole 1' to assist in reverse-sequence endoscopic nipple-sparing mastectomy combined with direct-to-implant breast reconstruction
  Interventions: Procedure: HUAXI hole 1
- Control group (No Intervention): Don't use 'HUAXI hole 1' to assist in reverse-sequence endoscopic nipple-sparing mastectomy combined with direct-to-implant breast reconstruction

INTERVENTIONS:
Procedure: HUAXI hole 1 — A small incision of 2mm is made at the junction of the upper outer edge of the areola and the skin, through which the scalpel is placed to assist in the resection of breast glands in reverse-sequence nipple-sparing mastectomy and direct-to-implant breast reconstruction.
  Arms: HH-01 group

SUMMARY:
This study is a multicenter, open-label, randomized controlled trial. It will prospectively compare outcomes between patients undergoing reverse-sequence endoscopic NSM (R-E-NSM) with direct-to-implant breast reconstruction (DIBR) with the "HUAXI Hole 1" versus without the "HUAXI Hole 1". The study aims to evaluate differences in operative efficiency, surgical safety, postoperative aesthetics, and oncological safety between the two groups.

DETAILED DESCRIPTION:
Conventional open nipple-sparing mastectomy (NSM) often results in significant surgical scarring, which is detrimental to the aesthetic outcome of the breast and the patient's psychosocial well-being. Meanwhile, endoscopic NSM has been reported to achieve favorable aesthetic outcomes and surgical safety. However, traditional endoscopic NSM has high technical difficulty and low surgical efficiency.

Our team has developed an innovative reverse-sequence endoscopic NSM (R-E-NSM) with direct-to-implant breast reconstruction (DIBR) following extensive research and clinical practice. This pioneering technique leverages the expansive force of gas to form a universal retractor. It employs an innovative reverse dissection sequence from deep to superficial layers, which retains the advantages of traditional endoscopic NSM while significantly improving operative efficiency. However, gland resection in the lower and inner quadrant of the breast remains technically challenging due to the long working distance and complex manipulation, often resulting in prolonged operative time and risks of incomplete gland resection.

To address these limitations, the West China Hospital team developed the "HUAXI Hole 1" technique-a 2-mm auxiliary incision at the superolateral edge of the areola, through which the electric scalpel is inserted to assist the gland resection. It can significantly reduce interference between instruments caused by the transaxillary single-incision approach and facilitate complete gland resection, which may contribute to improved surgical efficiency, surgical safety, and oncologic safety with the aesthetic advantages of the endoscopic technique. However, some researchers are concerned about the risks, such as nipple and areola complex (NAC) ischemia/necrosis, incision dehiscence, and surgical site infection. The prospective clinical evidence validating its efficacy and safety is currently lacking.

Therefore, this national multicenter, open-label, randomized controlled trial will prospectively compare outcomes between patients undergoing reverse-sequence endoscopic NSM (R-E-NSM) with direct-to-implant breast reconstruction (DIBR) with the "HUAXI Hole 1" versus without the "HUAXI Hole 1". The study aims to evaluate differences in operative efficiency, surgical safety, postoperative aesthetics, and oncological safety between the two groups.

ELIGIBILITY:
Inclusion criteria:

* Female patients aged 18-70 years (inclusive18 and 70 years);
* Patients eligible for unilateral or bilateral reverse-sequence endoscopic nipple-sparing mastectomy with immediate implant-based breast reconstruction, with concurrent contralateral endoscopic augmentation mammoplasty permitted;
* Patients with preoperative pathological confirmation of non-specialized breast cancer (e.g., ductal carcinoma in situ, invasive ductal carcinoma, invasive lobular carcinoma) or eligibility for prophylactic mastectomy;
* For non-specialized breast cancer patients, preoperative tumor size ≤5 cm (post-neoadjuvant chemotherapy if applicable), and no clinical or imaging evidence of invasion to the nipple, skin, subcutaneous fat, chest wall (referring to the bony thorax and intercostal muscles, excluding the pectoralis major and minor muscles) or distant metastasis preoperatively;
* Patients volunteered to provide informed consent.

Exclusion criteria:

* History of open breast surgery within 1 year before this procedure (excluding minimally invasive vacuum-assisted biopsy);
* Breast cancer diagnosed during pregnancy or lactation;
* Subnipple-plane scarring with radiotherapy;
* Metastatic breast cancer (M1);
* Severe comorbidities precluding general anesthesia or surgery;
* BMI ≥40 kg/m²;
* HbA1c >7.5%;
* Immunodeficiency;
* Active smoking with ≥20 cigarettes per day
* Patients with concurrent participation in conflicting clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative time | Immediate postoperative
  Overall operation time (minute) from skin incision to complete closure of incision, including breast cancer operations, lymph node surgery, and breast reconstructions.

SECONDARY OUTCOMES:
Complications | Immediate postoperative, within 3-month postoperative, and within 1-year postoperative
  Skin flap thermal injury, skin flap ischemia/necrosis, nipple and areola complex(NAC) ischemia/necrosis, surgical site infection, incision dehiscence, surgical site bleeding or hematoma, seroma needing repeated aspiration or drain reinsertion, capsular contracture, prosthesis outline appearance, rippling, implant displacement, implant loss, readmission
Aesthetic outcome evaluation--BREAST-Q scores | Preoperative (baseline), 3-month postoperative, and 2-year postoperative
  The Satisfaction with Breasts module of BREAST-Q questionnaire is utilized to assess patient-reported aesthetic outcomes. Transformed scores range from 0 to 100, with higher scores indicating better outcomes. Both raw questionnaire scores and standardized transformed scores will be documented, along with pre- to postoperative differences in transformed scores
Aesthetic outcome evaluation--Harris score | 3-month postoperative and 2-year postoperative
  The Harris score was used to record the subjective judgment of symmetry of the reconstructed breast compared to the contralateral breast. The results were categorized as excellent (treated breast nearly identical to untreated breast), good (treated breast slightly different than untreated), fair (treated breast clearly different than untreated), and poor (treated breast seriously distorted).
Aesthetic outcome evaluation--Ueda score | 3-month postoperative and 2-year postoperative
  Doctor-reported aesthetic outcomes will be evaluated by three professional breast surgeons using the Ueda scale, based on postoperative photographs. Scores range from 0 to 10 points, with higher values indicating better results. The categorized as follows: Excellent (≥9 points), Good (7-8 points), Fair (5-6 points), Poor (≤4 points). Both raw scores and categorizations will be documented
Quality of Life--BREAST-Q scores | Preoperative (baseline), 3-month postoperative, and 2-year postoperative
  The Psychosocial Well-Being, Sexual Well-Being, and Physical Well-Being of the Chest modules of BREAST-Q questionnaire are used to evaluate quality of life (QoL) outcomes. Transformed scores range from 0 to 100, with higher values indicating better outcomes. Both raw questionnaire scores and standardized transformed scores will be recorded, along with pre- to postoperative differences in transformed scores
Surgical margin involvement | 2-3 weeks postoperative after paraffin-embedded pathological report available
  Surgical margin involvement was defined as ink on tumor on postoperative paraffin-embedded pathological examination
Resection mastectomy weight | Immediate postoperative
  Mean mastectomy weight (g)
Local Recurrence-Free Survival(LRFS) | 2-year postoperative and 5-year postoperative
  The time interval from initiation of treatment to the first recurrence at the primary tumor site.If local recurrence appears, record the time and location of recurrence
Disease-Free Survival(DFS) | 2-year postoperative and 5-year postoperative
  The period from treatment initiation to any disease recurrence (local, regional, or distant) or death.If above event appears, record the time and disease location.
Overall Survival(OS) | 2-year postoperative and 5-year postoperative
  The time from treatment initiation (or diagnosis) to death from any cause. If death appears, record the time and reason.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Anyang City Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The Affiliated Hospital of lnner Mongolia Medical University, Hohhot, Inner Mongolia
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Taiyuan Central Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Fourth People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China hospital of Sichuan University, Chengdu, Sichuan
  - West China School of Public Health and West China Fourth Hospital, Sichuan University, Chengdu, Sichuan
  - West China Tianfu Hospital, Chengdu, Sichuan
  - Deyang People's Hospital, Deyang, Sichuan
  - Mianyang Hospital of Traditional Chinese Medicine, Mianyang, Sichuan
  - The People's Hospital of Dazu, Chongqing, Chongqing

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data via the request portal. All IPD requests should be emailed to Dr. Zhenggui Du, the general project leader, and will be evaluated by Dr. Du and the head of the collaborating organization to decide whether to approve.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of relevant research outputs, such as academic papers and books.
Access Criteria: When a request has been approved, the investigator will provide access to the de-identified individual patient-level data in the data management platform (Electronic Data Capture, EDC). A signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing the requested information. Additionally, all users will need to accept the terms and conditions of the data management platform to gain access.
URL: https://dct.meddb.cn/login_index

REFERENCES:
- [Background] Ho WS, Ying SY, Chan AC. Endoscopic-assisted subcutaneous mastectomy and axillary dissection with immediate mammary prosthesis reconstruction for early breast cancer. Surg Endosc. 2002 Feb;16(2):302-6. doi: 10.1007/s004640000203. Epub 2001 Nov 16. PMID 11967683
- [Background] Yang H, Liang F, Xie Y, Qiu M, Du Z. Single axillary incision reverse-order endoscopic nipple/skin-sparing mastectomy followed by subpectoral implant-based breast reconstruction: Technique, clinical outcomes, and aesthetic results from 88 preliminary procedures. Surgery. 2023 Sep;174(3):464-472. doi: 10.1016/j.surg.2023.05.037. Epub 2023 Jul 7. PMID 37422354
- [Background] Lai HW, Lin SL, Chen ST, Kuok KM, Chen SL, Lin YL, Chen DR, Kuo SJ. Single-Axillary-Incision Endoscopic-Assisted Hybrid Technique for Nipple-Sparing Mastectomy: Technique, Preliminary Results, and Patient-Reported Cosmetic Outcome from Preliminary 50 Procedures. Ann Surg Oncol. 2018 May;25(5):1340-1349. doi: 10.1245/s10434-018-6383-z. Epub 2018 Feb 26. PMID 29484564
- [Background] Zhou J, Xie Y, Liang F, Feng Y, Yang H, Qiu M, Zhang Q, Chung K, Dai H, Liu Y, Liang P, Du Z. A novel technique of reverse-sequence endoscopic nipple-sparing mastectomy with direct-to-implant breast reconstruction: medium-term oncological safety outcomes and feasibility of 24-h discharge for breast cancer patients. Int J Surg. 2024 Apr 1;110(4):2243-2252. doi: 10.1097/JS9.0000000000001134. PMID 38348883
- [Background] Qiu M, Liang F, Xie Y, Yang H, Zhang Q, Zhong J, Dai H, Du Z. Clinical Outcomes of Transaxillary Reverse-Sequence Endoscopic Nipple-Sparing Mastectomy and Direct-to-Implant Prepectoral Breast Reconstruction: A Prospective Study of Initial 68 Procedures. Ann Surg Oncol. 2024 Apr;31(4):2777-2785. doi: 10.1245/s10434-023-14687-7. Epub 2024 Feb 9. PMID 38334846
- [Background] Feng Y, Xie Y, Liang F, Zhou J, Yang H, Qiu M, Zhang Q, Liu Y, Liang P, Du Z. Twenty-four-hour discharge of patients after endoscopic nipple-sparing mastectomy and direct-to-implant breast reconstruction: safety and aesthetic outcomes from a prospective cohort study. Br J Surg. 2024 Jan 3;111(1):znad356. doi: 10.1093/bjs/znad356. No abstract available. PMID 37991082
- [Background] Lai HW, Chen DR, Liu LC, Chen ST, Kuo YL, Lin SL, Wu YC, Huang TC, Hung CS, Lin YJ, Tseng HS, Mok CW, Cheng FT. Robotic Versus Conventional or Endoscopic-assisted Nipple-sparing Mastectomy and Immediate Prosthesis Breast Reconstruction in the Management of Breast Cancer: A Prospectively Designed Multicenter Trial Comparing Clinical Outcomes, Medical Cost, and Patient-reported Outcomes (RCENSM-P). Ann Surg. 2024 Jan 1;279(1):138-146. doi: 10.1097/SLA.0000000000005924. Epub 2023 May 25. PMID 37226826
- [Background] Kim JH, Ryu JM, Bae SJ, Ko BS, Choi JE, Kim KS, Cha C, Choi YJ, Lee HY, Nam SE, Kim Z, Kang YJ, Lee MH, Lee JE, Park E, Shin HJ, Kim MK, Choi HJ, Kwon SU, Son NH, Park HS, Lee J; Korea Robot-endoscopy Minimal Access Breast Surgery Study Group. Minimal Access vs Conventional Nipple-Sparing Mastectomy. JAMA Surg. 2024 Oct 1;159(10):1177-1186. doi: 10.1001/jamasurg.2024.2977. PMID 39141399